CLINICAL TRIAL: NCT07352618
Title: "Effect of Omega-3 Supplementation as Add on Therapy on Glycemic Control and Lipid Profile in Type2 Diabetes Mellitus: A Randomized, Double-Blind, Placebo-Controlled Trial"
Brief Title: "Effect of Omega-3 Supplementation as Add on Therapy on Glycemic Control and Lipid Profile in Type2 Diabetes Mellitus."
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Bangladesh Medical University (Other)
Responsible Party: Principal Investigator, Dr. Toufique Tania Prity, Resident, Bangladesh Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BMU/2025/10266
Record Dates: First submitted 2026-01-12; First posted 2026-01-20 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-07

CONDITIONS: Type2 Diabetes Mellitus
MeSH Terms: interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Omega-3, (Experimental): Participant received Cap Omega-3 1gm orally twice daily for 12 weeks
  Interventions: Dietary Supplement: Omega-3 Fatty Acids
- Placebo (Placebo Comparator): Participants received Omega-3 placebo capsule matching Omega-3 orally twice daily for 12 weeks
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Omega-3 Fatty Acids — Participants received Omega-3 1gm capsule orally twice daily for 12 weeks
  Arms: Omega-3,
Dietary Supplement: placebo — Participants received Omega-3 placebo capsule twice daily for 12 weeks
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if Omega-3 works to control glycemic status, improve lipid profile in Type2 Diabetic patients. It will also learn about the safety of drug Omega-3. The main questions it aims to answer are:

Does drug Omega-3 control glycemic status, improve lipid profile in Type2 Diabetic patients? What medical problems do participants have when taking drug Omega-3? Researchers will compare Omega-3 to a placebo(a look-alike substance that contains no drug)to see if Omega-3 works to treat Type 2 Diabetic patients.

Participants will take Omega-3 or a placebo twice daily for 12 weeks. Baseline and 12 weeks after FPG, HbA1c,Serum Lipid profile, Omega-3 level will be monitored.

DETAILED DESCRIPTION:
Diabetes Mellitus is a common endocrine disorder. T2DM is characterized by polyuria, polydipsia, polyphagia. It affects both men and women. T2DM is strongly associated with impaired insulin sensitivity, insulin resistance, dyslipidaemia, hypertension, and central obesity. Omega-3 polyunsaturated fatty acid has been shown to exert beneficial effect on lipid metabolism and insulin sensitivity.

Aim of the study: We aimed to evaluate the effect of Omega-3 supplementation as add on therapy on glycemic control and lipid profile in Type 2 diabetes mellitus patients.

Methodology: This research will be a single center study, utilizing a double-blind, randomized placebo-controlled trial design. A total of 66 men and women, with diagnosed T2DM, age range from 25-75 years will randomly be assigned to receive either Omega-3 supplementation or placebo for 12 weeks. Biochemical and anthropometric measurements, including Fasting plasma glucose, HbA1c, lipid profile, blood pressure, BMI, waist-hip ratio and waist-to-height ratio will be assessed at baseline and post-treatment. Follow-up assessments will be conducted after supplementation for 12 weeks to evaluate the sustainability of biochemical changes. For independent samples; t-test will be utilized to analyze the average differences in metabolic biomarker levels between the group receiving Omega-3 supplements and the group receiving a placebo. The Chi-square test or Fisher's exact test will be employed to compare the percentage of participants may show a significant change in metabolic biomarker in the group that received Omega-3 versus the group that received a placebo.

Pearson or Spearman correlation tests will be used to explore any relationships between baseline Omega-3 levels and FPG, HbA1c and lipid profile levels, as well as between the change in Omega-3 levels and the change in FPG, HbA1c and lipid profile levels.

Conclusion: Combining Omega-3 supplementation with the conventional treatment could potentially have a substantial impact on lipid profile and glycemic control in patients with T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Age above 25 years up to 75 years
* Old and newly diagnosed case of Type2 DM.
* Patient receiving conventional diabetic treatment like OAD or insulin or both
* Patient may have altered lipid profile or not
* Both male and female patient
* Patient's HbA1c level within 8.0%

Exclusion Criteria:

* Pregnancy and lactating mother.
* History of known Type1 diabetes mellitus, secondary diabetes, drug induced diabetes, drugs interfering body weight.
* Patient with acute illness, liver disease, psychiatric disorder
* Patients receiving Omega-3 supplementation within the last three months.
* Known allergy to fish oil or Omega-3 supplements.

Ages: 25 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Changes in lipid profile | 12 weeks
  (triglycerides, HDL-Cholesterol)
Change in Plasma Omega-3 level | 12 weeks
  changes in plasma DHA and EPA conc
Change in HbA1c | 12 weeks
Improvement of Fasting Plasma Glucose | 12 weeks

SECONDARY OUTCOMES:
Change in Blood Pressure (Systolic and Diastolic Blood Pressure) | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Bangladesh Medical University, Dhaka, Bangladesh